CLINICAL TRIAL: NCT02103088
Title: PROCAN: Sexual and Urological Rehabilitation to Men Operated for Prostate Cancer and Their Partners: A Randomized Controlled Intervention Study
Brief Title: Sexual and Urological Rehabilitation to Men Operated for Prostate Cancer and Their Partners
Acronym: PROCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: The Capital Region Research Foundation for Health Research Denmark (Unknown); Rigshospitalet, Denmark (Other); Clinic for Sexology and Center for Psychiatry Copenhagen Denmark (Unknown)
Responsible Party: Principal Investigator, Christoffer Johansen, MD, PhD, Dr. Med.Sci, Head of Unit, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROCAN
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Intervention; Rehabilitation; Couple; Sexology; Urology; Late effects
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sexual and urological intervention (Experimental): Standard care and the PROCAN intervention consisting of i) DVD instruction in pelvic floor muscle training ii) group instructions in pelvic floor muscle training by physiotherapist including three individually follow-up and ii) up to six couple sessions performed by a sexual nurse counselor.
  Interventions: Behavioral: Sexual and urological intervention
- Control (No Intervention): Standard care consists of:systematic offer of medical treatment for erectile dysfunction, if not contra indicated. The medical treatment will consist of either daily treatment with Cialis 5 mg or phosphodiesterase type 5 inhibitor on demand before sexual activity. Alternatively use of alprostadil as either urethral pin or penile injection. Furthermore standard treatments include preoperative instruction in pelvic floor muscle training, regular outpatient visits and possible referral to rehabilitation in accordance with the rules that apply to the Danish Health legislations. In case of prolonged incontinence the patients may on request be referred to a private practicing physiotherapist.

INTERVENTIONS:
Behavioral: Sexual and urological intervention — Sexual and urological intervention consisting of: i) DVD instruction in pelvic floor muscle training ii) group instructions in pelvic floor muscle training by physiotherapist including three individually follow-up and ii) up to six couple sessions performed by a sexual nurse counselor.
  Arms: Sexual and urological intervention

SUMMARY:
Today prostate cancer (PC) treatment with curative intent is primarily surgical removal of the prostate gland (prostatectomy) which may be associated with immediate and long lasting erectile dysfunction and decline in urinary function. Besides these physical late effects patients operated for PC have a twofold increased risk for depression up to ten years after the diagnosis. To reduce these late effects affecting both patient and partner the investigators have developed a sexual and urological intervention (PROCAN). The intervention is based on epidemiological data, evidence from previous clinical trials, a feasibility study and qualitative explorations among PC patients and partners. The investigators hereby suggest the conduction of a randomized controlled trial to test the effect of the PROCAN intervention on urological and sexual dysfunction, couples adjustment and quality of life. Results of the proposed trial may provide clinicians and decision makers with the evidence needed to optimize rehabilitation after PC.

DETAILED DESCRIPTION:
Although the potential negative impact of prostate cancer on sexual and urological function is well documented there is no evidence based and standardized rehabilitation offer available for Danish couples affected by prostate cancer. This study proposal is based on a thorough literature review on PC treatment and late effects and interventions targeting sexual and urological late effects and a qualitative study including interviews with 6 couples affected by PC. The literature review showed that; medical treatment is effective for the treatment of erectile dysfunction, psychosocial intervention may ease sexual problems secondary to operation for prostate cancer and sexual counseling may improve compliance with medical treatment of erectile dysfunction. In regard to treatment of urological dysfunction studies showed that the effect of pelvic floor muscle training is enhanced by follow-up instructions by physiotherapist. Our interview study among patients operated for prostate cancer and their partners indicated a general need and demand for professional help to discuss the changed sexual life. Also studies have shown that health professionals find it difficult to discuss sexual problems with the patients. Medical treatment for erectile dysfunction is prescribed to patients operated for prostate cancer, however the treatment is not offered systematically in all hospitals and furthermore the drugs are sold on the internet.In view of this knowledge we determine that there is a need for studies which include patients systematically offered medical treatment for erectile dysfunction and further is offered sexual counseling and thus focusing on: i) treatment of physical, psychological and social aspects of sexual dysfunction ii) improvement of compliance with the medical treatment for erectile dysfunction and iii) reducing barriers among patients and health professionals for resolving sexual problems secondary to operation for prostate cancer.

The purpose of the PROCAN study is in a randomized design to test the effect of a theory based intervention on sexual and urological dysfunctions secondary to operation for prostate cancer. The PROCAN intervention consists of: i) Digital Video Disc (DVD) instruction in pelvic floor muscle training ii) group instructions in pelvic floor muscle training by physiotherapist including up to three individually follow-up and ii) up to six couple sessions performed by a sexual nurse counselor. The intervention is based on social and cognitive behavioral techniques and techniques derived from sexual therapy and counseling with a psycho-educational approach, in which sexuality is defined as a multidimensional construct involving biological, psychological and social aspects. The intervention is documented and developed in collaboration with urologists, physiotherapists and sexologists. The investigators will enroll patients and partners from the Urological Department Rigshospitalet and randomize 160 couples. Patients and partners will be randomized (1:1) to standard care plus the PROCAN intervention and to standard care (control Group). The investigators hypothesize that the PROCAN intervention will:

* Improve urological and sexual functioning among prostate cancer patients and sexual function and satisfaction among patients and female partners
* Improve the dyadic adjustment and the overall quality of life in prostate cancer patients and their partners
* Reduce the prevalence of depression and anxiety in patients and their partners

ELIGIBILITY:
Inclusion Criteria: Patients operated for primary prostate cancer with open or robot-assisted surgery using nerve sparring or non-nerve sparring technique living with a female partner and reported being sexually active before the operation.

Exclusion Criteria:Patients with other cancers (except non-melanoma skin cancer) within 5 years, major psychiatric disorder, abuse of alcohol or drugs, dementia, e.g. Alzheimer's disease and patients, who do not understand or speak Danish. Patients, who reported not being sexually active before the operation and partners who do not understand or speak Danish.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05; Primary Completion 2019-01 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Erectile function measured by the International Index of Erectile Function (IIEF-15) | Baseline, 8 months and 12 months
  To investigate the change in erectile function among patients in intervention- and the control group from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group

SECONDARY OUTCOMES:
Sexual satisfaction measured by IIEF-15 | Baseline, 8 and 12 months
  To investigate the change in sexual satisfaction among patients from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Female sexual satisfaction measured by The Female Sexual Function Index (FSFI) | Baseline, 8 and 12 months
  To investigate the change in sexual satisfaction among female partners from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Female Sexual Distress measured by the Female Sexual Distress Scale (FSDS) | Baseline, 8 and 12 months
  To investigate the change in female sexual distress from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Urological function measured by The Expanded Prostate Cancer Composite Index (EPIC-26) | Baseline, 8 and 12 months
  To investigate the change in urological function among patients from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Marital function measured by The Dyadic Adjustment Scale (DAS) | Baseline, 8 and 12 months
  To investigate the change in marital function among patients and partners from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Health related quality of life measured by The Short Form Health Survey (SF-36) | Baseline, 8 and 12 months
  To investigate the change in health related quality of life among patients and partners from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Anxiety measured by The Symptom Check List (SCL-92) | Baseline, 8 and 12 months
  To investigate the change in anxiety among patients and partners from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group
Depression measured by The Major Depression Inventory (MDI) | Baseline, 8 and 12 months
  To investigate the change in depressive symptoms among patients and partners partners from baseline to 8 and 12 months follow up and the difference in change between intervention - and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, PhD, Dr. Med, Principal Investigator — Danish Cancer Society; Randi V. Karlsen, RN, MEd, Principal Investigator — Danish Cancer Society
Locations (1):
- Department of Urology, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark